CLINICAL TRIAL: NCT00884338
Title: Evaluation of the Cognitive Function of Patients After Stem Cell Transplantation
Brief Title: Cognitive Function After Stem Cell Transplantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Dr. Fernando Dimeo, Charite Universitätsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA4/028/09
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Fatigue; Cognitive Impairment; Stem Cell Transplantation
Keywords: Fatigue; Cancer; Cognitive impairment; Exercise; Sport; Peripheral blood stem cell transplantation; High-dose chemotherapy
MeSH Terms: conditions — Fatigue; Cognitive Dysfunction; Neoplasms; Motor Activity | interventions — Counseling

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Other: Endurance exercise
- Control group (Active Comparator)
  Interventions: Other: Counseling

INTERVENTIONS:
Other: Endurance exercise — The patients will carry out an endurance exercise program consisting of walking on a treadmill for 30 to 40 minutes at a speed corresponding to 80% of the maximum heart rate
  Arms: Exercise
Other: Counseling — Counseling about exercise and behavioural techniques to reduce fatigue
  Arms: Control group

SUMMARY:
The trial will evaluate the effects of an exercise program on the physical and cognitive performance of patients with hematological neoplastic diseases after high dose chemotherapy with stem cell support.

DETAILED DESCRIPTION:
Patients (n = 60) will be randomized to an exercise or a control group. The randomization will be stratified for allogeneic or autologous blood stem cell transplantation. Patients in the exercise group will carry out an endurance training consisting of walking on a treadmill at a speed corresponding to 80% of the maximum heart rate. The exercise program will be carried out 3 times weekly for 8 weeks. Patients in the control group will receive counseling about exercise and behavioural techniques to reduce fatigue, but they will not participate at a structured exercise program. Physical performance (VO2max), cognitive function, mood and quality of life will be evaluated at recruitment and after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70
* Hematological neoplastic disease
* Treatment with high-dose chemotherapy with peripheral blood stem cell transplantation in the previous 3 years
* Karnofsky-Index > 80%
* Ability to understand German

Exclusion Criteria:

* Cardiorespiratory, metabolic, inflammatory or osteoarticular diseases which can be aggravated by exercise
* Psychosis
* Organic brain damage
* Dementia
* PBSCT in the previous 6 weeks
* Pathological stress test at admission

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-08 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
VO2max | Recruitment and after 8 weeks

SECONDARY OUTCOMES:
Cognitive status, mood, quality of life | At recruitment and after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Dimeo, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany